CLINICAL TRIAL: NCT02594774
Title: Efficacy of Osteopathic Treatment in Function Abdominal Pain in Children and Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Oscar Garcia Algar, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/6312/I
Record Dates: First submitted 2015-10-30; First posted 2015-11-03 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteopathic treatment (Experimental): Manipulative osteopathy (and standard medical treatment)
  Interventions: Other: Manipulative osteopathy
- Standard medical treatment (No Intervention): Standard medical treatment

INTERVENTIONS:
Other: Manipulative osteopathy — Osteopathic treatment (BMT) which works on the influence on the pressure distribution in the (especially abdominal) body cavities and consequently on the viscera contained therein, proper arterial supply and venous and limphatic drainage.
  Arms: Osteopathic treatment

SUMMARY:
The objective is to evaluate the efficacy of osteopathic treatment as an adjunct to standard medical treatment in reducing child functional abdominal pain.

A convenience sample that includes no more than 30 patients per study group (n = 60) are being recruited. As an exploratory study the investigators did not proceed to make any sample size calculation.

This is a comparative study of two quasi-experimental interventions (standard treatment vs. standard treatment + Osteopathy).

This will be a single-blind trial where only the evaluator will be blinded. The principal outcome will be pain measured by a visual analog scale. A version with more appropriate pictograms for pediatric patients is used. Measurements will be taken at baseline (baseline measurements) at 4, 8 weeks (the duration of interventions) and 6 months post-study.

DETAILED DESCRIPTION:
Although the functional or structural disease can be identified by physicians and sometimes cured by medical technology, non-structural or functional symptoms, those without an identified organic cause and associated with a high rate of response to placebo are yet enigmatic and less susceptible to explanation or effective treatment.

Often considered as non-pathological, there are physiological and sociocultural factors, nociceptive, psychic that expand the perception of these symptoms which are experienced as serious, problematic and threatening with the consequent impact on daily activities. Although it represents the most frequent cause of consultation in the specialty of Pediatric Gastroenterology there is currently no drug therapy that has demonstrated its effectiveness.

In these cases, unnecessary diagnostic studies can be performed to find an organic cause, resulting in increased health care costs and possibly in an inappropriate patient care. These types of beliefs and behaviors can delegitimize the DFG and the suffering of these patients.

There are studies that say that 35% of patients suffering from irritable bowel syndrome (no organic cause but if organic effect) use complementary therapies, but in the absence of clinical trials, it is emphasized the need for more controlled studies to advise and / or direct the patient from the medical community to which of these therapies could be more adequate.

According to the General Osteopathic Council (UK) and the Osteopathic International Alliance (OIA), Osteopathy is a health profession that is dedicated to the diagnosis, treatment and prevention of problems of the musculoskeletal and its effects on the nervous system and global health. It is based on the theory that well-being depends on a good relationship between the skeleton, muscles, ligaments and connective tissue. The lack of this good relationship can lead to symptoms and musculoskeletal problems but also visceral. Health is seen as a complex process involving all parts and systems of the body. Palpatory techniques are used to diagnose dysfunction and physical manipulation is used to improve the functioning of joints, relax muscle tension, promote the innervation and blood supply to tissues and help the healing mechanisms of the body.

There are studies in the field of Osteopathy evaluating the efficacy of this approach in different intestinal dysfunctions and diseases. Da Silva et al demonstrated the usefulness of increasing the pressure of the lower esophageal sphincter in the osteopathic approach in patients with gastroesophageal reflux. Attali et al suggested that visceral osteopathy improves short and long term bloating and rectal sensitivity in patients with irritable bowel syndrome. Florance et al reported improvements in quality of life and symptomatic improvement in patients with irritable colon with a pilot study and Piche et al showed reduced severity of symptoms associated with irritable bowel in patients with Crohn's disease in remission. The positive effect of osteopathic treatment in the management of symptoms caused by irritable bowel syndrome was confirmed in a couple of systematic reviews recently published.

However, all these studies were performed with adult patients. On a pediatric level, most of the literature focuses on infant colic. The most notable reference is the Cochrane review in 2012 in which several manipulative therapies are evaluated in the. One of the weaknesses identified in this review is that parents entrusted to objectify the improvements were not blinded. This defect is corrected in a subsequent study in the chiropractor field. The effectiveness of osteopathic treatment for infantile colic has also been studied but always with small samples or methodological flaws. An example is the study by Hayden et al. Silva et al which shows that the use of physical therapy (muscle exercises, breathing and abdominal massage) is effective in pediatric chronic constipation with defecation increasing frequency.

The scientific evidence regarding the effectiveness of osteopathic treatment on digestive disorders in both adults and pediatric patients is limited and constrained. At the same time, there are no studies in the pediatric setting on approach through manual therapy in abdominal painful functional disorders.

OBJECTIVES

* Primary Objective: To evaluate the efficacy of osteopathic treatment as an adjunct to standard medical treatment in reducing child functional abdominal pain.
* Secondary Objectives: To evaluate the influence of osteopathic treatment in children and adolescents with functional abdominal pain related to absenteeism, the number of emergency room visits, quality of life and the need for rescue medication. The potential adverse effects were recorded.

METHODS

1. Design: Controlled clinical trial single-blind
2. Site where the study is conducted:

   Participants will be recruited in the following pediatric services where medical intervention is carried out:

   Hospital del Mar de Barcelona Hospital Sant Joan de Déu de Barcelona Participants in the experimental group (standard medical treatment + osteopathic treatment) will be referred to d'Osteopathy Clinic of Barcelona for the realization of osteopathic treatment.
3. Sample:

   A convenience sample that includes no more than 30 patients per study group (n = 60) are being recruited. As an exploratory study the investigators did not proceed to make any sample size calculation.
4. Eligibility Criteria:

   Inclusion criteria: The sample consists in patients of school age (6-16 years old) diagnosed with functional abdominal pain (Functional Abdominal Pain-Related Disorders) according to the diagnostic criteria for functional gastrointestinal disorders ROME guide III.

   Exclusion criteria: Patients diagnosed with digestive disease, patients who have or are receiving medical aids and patients who are not studying physical treatments.
5. Randomization:

This is a comparative study of two quasi-experimental interventions (standard treatment vs. standard treatment + Osteopathy). The allocation of the patients in each group will be held (after obtaining informed consent) through a system of randomization plus a matching system. Patients who meet the eligibility criteria will be randomized to receive one or other intervention in the first instance.

This allocation to the study groups will be marked and induce the pairing ("matching") to a new subject of study that meets the same characteristics as the previously randomized. To do this, during random award, 3 specific characteristics of the subjects will be recorded:

1. age (from 6 years to 10 years and 11 to 16 years)
2. sex
3. type of functional abdominal pain and severity (ROME III). When a new patient with the same characteristics previously patients randomized to a study group, it will be assigned paired to form another study group without going through a randomization process again.

With this design the investigators intend to balance study groups given that the investigators will have a small sample and with a pragmatic inclusion.

f) Masking: This will be a single-blind trial where only the evaluator will be blinded. The characteristics of the studied intervention is not possible to mask nor the therapist or the patient.

g) Interventions:

* Standard medical treatment: organic cause has to be discarded through complementary examinations, depending on the symptoms of each patient. Subsequently, the appropriate standard pharmacological treatment for each type of functional abdominal pain will be applied:
* Functional dyspepsia: proton-pump inhibitor omeprazole 1 mg / kg / day vo
* Abdominal migraine -Treatment: sumatriptan 50 mg PO
* Functional abdominal pain: antispasmodics
* Irritable colon: methylcellulose + antispasmodics

  * There are few studies to define the precise standard treatment of functional abdominal pain
* Osteopathic treatment (BMT) description collecting the items of the interventions guide report tidier. The TMO is a 100% manual intervention applied individually with direct contact between therapist and patient. For this study 5 sessions are set with a fortnightly interval between sessions and lasts between 45 and 60 'each (total 2 months of treatment).

Both on the first visit and other physical examination prior to treatment consisting will be held:

i. Quadrant abdominal palpation ii. Rating excursion tone and respiratory and pelvic diaphragm iii. Palpation and mobility tests of the spine (especially high thoracic and lumbar segments) iv. Test listening in skull base and cranial sacral following the model of William G. Sutherland.

Scanning is performed to detect the presence of somatic dysfunction (DS). The term DS is part of osteopathic terminology and is defined as "alterations in the function of the components related to the somatic system: skeletal structures, joint and myofascial and vascular elements, neural and lymphatic related".

The scan results will determine the treatment that will be adapted to each particular case but within the framework and following techniques:

* See the complete description of the techniques Glossary of Osteopathic Terminology, 2011.

  1. Indirect Techniques for working the abdominal and pelvic diaphragm Objective: To work on the influence on the pressure distribution in the (especially abdominal) body cavities and consequently on the viscera contained therein, proper arterial supply and venous drainage and linfático.
* Osteopathic models to justify this approach and other related references. 2. Functional Techniques for visceral dysfunctions Objective: visceral relaxation techniques. Listen and treatment of visceral motility by functional techniques applied directly to the viscera and their supporting tissues
* Osteopathic models to justify this approach and other related references. 3. Direct Techniques (articulatory) and / or indirect spine dysfunctions 4. Treatment by cranial sacral approach to dysfunction and skull Objective: Work on visceral autonomic innervation (sympathetic and parasympathetic) to the different digestive organs in order to improve vascularization and function.

Who will perform the intervention ?:

A unique osteopath (DM) will carry out all interventions to avoid as far as possible biases among different therapists. DM is a Physiotherapist and Osteopath with over 10 years of clinical experience in both adults and pediatric patients. She is specialized in pediatric Osteopathy through postgraduate training.

Strategies to ensure adherence to treatment and co-interventions such as telephone reminder scheduled visits for osteopathic treatment. Special care will be taken to avoid co-interventions. To do so participants at baseline was duly informed through a special paragraph in the informed consent h) Outcomes:

* Principal outcome: Pain Measured by a visual analog scale. A version with more appropriate pictograms for pediatric patients is used. Measurements will be taken at baseline (baseline measurements) at 4, 8 weeks (the duration of interventions) and 6 months post-study
* Secondary outcomes:

  * Truancy: a record of truancy during the 6 months follow-up study
  * Number of visits to the emergency: a registry of emergency room visits during the 6 months follow-up study
  * Quality of life: Patients will fill out the form Kidscreen quality of life in its translation into Spanish (at the beginning and end of the study)
  * Calendar symptoms: Patients have to fill out a schedule of symptoms 6 months follow-up study with the following variables: days of onset of pain, pain intensity, pain location, triggers, associated symptoms and need taking rescue medication.
  * Adverse effects: a record of the adverse effects that might occur during the study

ELIGIBILITY:
Inclusion Criteria:

* Patients of school age (6-16 years old)
* Diagnosed with functional abdominal pain (Functional Abdominal Pain-Related Disorders) according to the diagnostic criteria for functional gastrointestinal disorders ROME guide III
* Signed informed consent

Exclusion Criteria:

* Patients diagnosed with digestive disease
* Patients who have or are receiving medical aids
* Patients who are not studying physical treatments
* Refusal to participate

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain (visual analog scale) | Baseline, 4 weeks, 8 weeks, 6 months
  Pain measurement through visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: CRISTINA MOLERA-BUSOMS, Principal Investigator — Hospital del Mar
Locations (1):
- Parc de Salut Mar, Barcelona, Spain

REFERENCES:
- [Background] Drossman DA. The functional gastrointestinal disorders and the Rome III process. Gastroenterology. 2006 Apr;130(5):1377-90. doi: 10.1053/j.gastro.2006.03.008. No abstract available. PMID 16678553
- [Background] Saps M, Biring HS, Pusatcioglu CK, Mintjens S, Rzeznikiewiz D. A comprehensive review of randomized placebo-controlled pharmacological clinical trials in children with functional abdominal pain disorders. J Pediatr Gastroenterol Nutr. 2015 May;60(5):645-53. doi: 10.1097/MPG.0000000000000718. PMID 25906454
- [Background] van Tilburg MA, Palsson OS, Levy RL, Feld AD, Turner MJ, Drossman DA, Whitehead WE. Complementary and alternative medicine use and cost in functional bowel disorders: a six month prospective study in a large HMO. BMC Complement Altern Med. 2008 Jul 24;8:46. doi: 10.1186/1472-6882-8-46. PMID 18652682
- [Background] Hussain Z, Quigley EM. Systematic review: Complementary and alternative medicine in the irritable bowel syndrome. Aliment Pharmacol Ther. 2006 Feb 15;23(4):465-71. doi: 10.1111/j.1365-2036.2006.02776.x. PMID 16441466
- [Background] Attali TV, Bouchoucha M, Benamouzig R. Treatment of refractory irritable bowel syndrome with visceral osteopathy: short-term and long-term results of a randomized trial. J Dig Dis. 2013 Dec;14(12):654-61. doi: 10.1111/1751-2980.12098. PMID 23981319
- [Background] Muller A, Franke H, Resch KL, Fryer G. Effectiveness of osteopathic manipulative therapy for managing symptoms of irritable bowel syndrome: a systematic review. J Am Osteopath Assoc. 2014 Jun;114(6):470-9. doi: 10.7556/jaoa.2014.098. PMID 24917634
- [Background] Dobson D, Lucassen PL, Miller JJ, Vlieger AM, Prescott P, Lewith G. Manipulative therapies for infantile colic. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD004796. doi: 10.1002/14651858.CD004796.pub2. PMID 23235617